CLINICAL TRIAL: NCT02559128
Title: The Role of Insulin Resistance in Patients With Heart Failure and Type 2 Diabetes
Acronym: CARMET2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Prof. Terezie Pelikanova, Prof. Terezie Pelikánová, MD.,PhD., Institute for Clinical and Experimental Medicine
Other Study IDs: G 15-06-02
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Insulin Resistance; Chronic Heart Failure
Keywords: Insulin Resistance; Chronic Heart Failure; Type 2 Diabetes; Endothelial Dysfunction
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- HF+T2D+: 40 patients with chronic HF and type 2 diabetes or prediabetes without previous pharmacological treatment
- HF+T2D-: 20 subjects with HF without T2D or prediabetes
- HF-T2D+: 20 subjects with T2D or prediabetes alone
- HF-T2D-: 20 healthy control volunteers

SUMMARY:
The purpose of this cross-sectional comparative 2x2 trial study is to compare the degree of insulin resistance, myocardial function and selected metabolic parameters and to explore the pathophysiological mechanisms by which insulin resistance is implicated in development of chronic heart failure (HF) in patients with type 2 diabetes and prediabetes (T2D).

Investigators hypothesize that patients with heart failure will be insulin-resistant and will display metabolic abnormalities as patients with diabetes.

DETAILED DESCRIPTION:
100 subjects in total, divided into four groups will be included: 40 patients with type 2 diabetes or prediabetes and chronic HF without previous pharmacological treatment (T2D+HF+), 20 subjects with HF without T2D (HF+T2D-), 20 subjects with T2D alone (HF-T2D+) and 20 healthy control volunteers (HF-T2D-).

All examinations will be done during a short admission at Diabetes Center (CD) in Institute for Clinical and Experimental Medicine (IKEM), always under comparable circumstances. All participants will undergo standardized selection of metabolic and cardiovascular tests.

Oxidative stress markers, selected cytokines, peptides and metabolites in blood and subcutaneous adipose tissue will be analyzed. Investigators assume that this project will bring new knowledge which will contribute to discovery of the mechanisms implicated in the development of heart failure in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

A. For group HF+T2D+

1. Chronic heart failure will be defined by the following criteria (all must be included):

   * diagnosis of HF known for at least 6 months
   * medical history of hospitalization for cardiac decompensation with need for parenteral therapy for congestion - X-ray findings or swelling of lower extremities
   * stable drug therapy at least 1 month
   * treatment with diuretics (thiazide or furosemide)
   * left ventricular ejection fraction (LVEF) below 50%
2. The presence of diabetes/prediabetes will be defined by:

   * diagnosis and treatment of type 2 diabetes in the medical history
   * or estimated screening blood sample: values of HbA1c (according to IFCC) ≥39 mmol/mol for prediabetes, ≥48 for diabetes and fasting plasma glucose level ≥5.6 mmol/l for prediabetes and ≥7 mmol/l for diabetes or ≥7.8 mmol/l for prediabetes and ≥11.1 mmol/l for diabetes according to oral glucose tolerance test (oGTT).
   * treatment of diabetes - by diet only
   * women and men aged 40-70 years
   * body mass index (kg/m2) in the range of 20-35
   * the range of HbA1c between 40-65 mmol/mol (IFCC)
   * signed informed consent

B.For group HF+T2D-

Chronic heart failure will be defined by the following criteria (all must be included):

* diagnosis of HF known for at least 6 months
* medical history of hospitalization for cardiac decompensation with need for parenteral therapy for congestion - X-ray findings or swelling of lower extremities
* stable drug therapy at least 1 month
* treatment with diuretics (thiazide or furosemide)
* LVEF below 50%
* no history of diabetes, HbA1c <39 mmol/mol (IFCC) and fasting plasma glucose level under 5.6 mmol/l
* women and men aged 40-70 years
* body mass index (kg/m2) in the range of 20-35
* signed informed consent

C.For group HF-T2D+

The presence of diabetes/prediabetes will be defined by:

* diagnosis and treatment of type 2 diabetes in the medical history
* or estimated screening blood sample: values of HbA1c (according to IFCC) ≥39 mmol/mol for prediabetes, ≥48 for diabetes and fasting plasma glucose level ≥5.6 mmol/l for prediabetes and ≥7 mmol/l for diabetes or ≥7.8 mmol/l for prediabetes and ≥11.1 mmol/l for diabetes according to oGTT
* treatment of diabetes - by diet only
* women and men aged 40-70 years
* body mass index (kg/m2) in the range of 20-35
* the range of HbA1c between 40-65 mmol/mol (IFCC)
* no history of acute or chronic heart disease
* signed informed consent

D.For group HF-T2D-

Absence of metabolic syndrome (not more than any two of the following symptoms):

* abdominal obesity - waist circumference in men> 102 cm, in women > 88 cm
* diagnosis and treatment of type 2 diabetes or raised fasting plasma glucose level (FPG> 5,6 mmol/l)
* raised blood pressure (BP): systolic BP > 130 mm Hg or diastolic BP >85 mm Hg, or treatment of previously diagnosed hypertension
* reduced HDL cholesterol in men < 1 mmol/l, in women < 1,3 mmol/l (or treatment)
* raised triglycerides > 1,7 mmol/l (or treatment)
* absence of chronic or acute cardiovascular disease
* women and men aged 40-70 years
* body mass index (kg/m2) in the range of 20-35
* signed informed consent

Exclusion Criteria groups (A+B+C+D):

* metabolic disease, including: 1 type diabetes, decompensated thyreopathy (Note: patients with hypothyroidism and stable substitution (the last 3 months) of normal thyrotropic-stimulating hormone levels may participate in the study)
* pregnancy (positive human chorionic gonadotropin test), breast feeding, trying to become pregnant
* clinically significant anemia with hemoglobin below 100 g/l
* renal insufficiency with estimated glomerular filtration under 0.7 ml/s
* atrial fibrillation
* alcoholism or drug use
* the presence of other medical condition, which occurs during physical examination, laboratory tests, ECG, including pulmonary, neurological or inflammatory disease, which would be considered by the examiner to distort the consistency of data

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 subjects in total, divided into four groups will be included: 40 patients with type 2 diabetes or prediabetes and chronic heart failure (HF+T2D+), 20 subjects with HF without T2D (HF+T2D-), 20 subjects with T2D alone (HF-T2D+) and 20 healthy control volunteers (HF-T2D-).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | At baseline
  Difference in glucose disposal rate and metabolic clearance rate of glucose measured by hyperinsulinemic euglycemic clamp
Heart function | At baseline
  Difference in left ventricular ejection fraction (LV EF), diastolic function (E/E´, left atrial volume) and ventriculi-vascular coupling measured by non-invasive estimation of end-systolic left ventricular (Ees) and arterial elastance (Ea) by single beat method measured by ECHO
Exercise capacity | At baseline
  Difference in peak oxygen consumption (peak VO2) and chronotropy index measured by symptom-limited bicycle spiroergometry

SECONDARY OUTCOMES:
Gut microbiota spectrum in stool and gut microbe generated trimethylamine N-oxide (TMAO) in plasma | At baseline
Endothelial function | Change in digital pulse amplitude tonometry from the basal state before the clamp and at the end f the measurement
  Change in endothelial function by acute artificial hyperinsulinemia measured by digital pulse tonometry during hyperinsulinemic euglycemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Terezie Pelikánová, Prof., MD, Principal Investigator — Diabetes Center, Institute of Clinical and Experimental Medicine, Prague, Czech Republic
Locations (1):
- Diabetes Center, Institute of Clinical and Experimental Medicine, Prague, Prague 4, Czechia